CLINICAL TRIAL: NCT05994365
Title: A Real-world Study of Anlotinib Hydrochloride Capsules in the Treatment of Locally Advanced or Metastatic Radioiodine-Refractory Differentiated Thyroid Carcinoma
Brief Title: Study of Anlotinib Hydrochloride Capsules in the Treatment of Locally Advanced or Metastatic Radioiodine-Refractory Differentiated Thyroid Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: A LOT-DTC-1
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anlotinib group: Anlotinib hydrochloride capsules: 12 mg once daily for 2 weeks, followed by a discontinuation of 1 week (21 days as a cycle)
  Interventions: Drug: Anlotinib Hydrochloride Capsule
- Observation group: Observation: prospectively and retrospectively collect data of patients who did not receive anlotinib hydrochloride capsules or similar small-molecule antivascular inhibitors.

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsule — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor that inhibits both tumor angiogenesis and tumor cell proliferation.
  Groups: Anlotinib group

SUMMARY:
The study aims to observe and investigate the efficacy and safety of Anlotinib capsules in patients with locally advanced or metastatic radioiodine-refractory differentiated thyroid carcinoma in the real world, and to summarize the treatment experience in a broad population.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in this study, sign the informed consent form and had good compliance;
* Aged 18 ~ 70 years old; Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0~1; more than 6 months of expected survival ;
* Histopathologically confirmed locally advanced or metastatic differentiated thyroid cancer, radiographically documented disease progression within 18 months of absence of radioactive iodine (RAI) therapy;
* Meet any of the following:

  1. Lesions were not iodine-avid: no RAI uptake was confirmed after RAI scan in the presence of a low-iodine diet, adequate thyroid stimulating hormone (TSH) elevation (≥ 30 mIU/L). The definition of no iodine uptake:

     1. no iodine uptake initially;
     2. exist of iodine uptake initially while lost subsequently;
     3. partially uptake;
     4. progression disease despite iodine uptake.
  2. The cumulative dose of RAI was ≥ 600 mCi or 22 GBq, with an interval of at least 3 months.
  3. Radiographically documented disease progression within 18 months of RAI therapy despite the presence of iodine-131 affinity at the time of RAI therapy;
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
* Major organ functions meet the following criteria within 7 days prior to treatment:

  1. Blood routine test criteria (14 days without blood transfusion):

     1. Hemoglobin (HB) ≥ 85 g/L;
     2. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
     3. Platelet (PLT) ≥ 80 × 10^9/L
  2. Biochemical tests need to meet the following criteria:

     1. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN);
     2. Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2 .5×ULN, ALT and AS if liver metastases T ≤ 5 ×ULN;
     3. Serum creatinine (Cr) ≤ 1 .5 ×ULN or creatinine clearance (CCr) ≥ 60 Ml/min;
* Females of childbearing potential should agree to use contraceptive measures (such as intrauterine device, contraceptives or condoms) during the study and within 6 months after the end of the study; have a negative serum or urine pregnancy test within 7 days before study enrollment and must be non-lactating patients; and males should agree to use contraceptive measures during the study and within 6 months after the end of the study period.

Exclusion Criteria:

* Comorbidities and medical history:

  1. A history of or concurrent with other malignancies within the past 3 years. Patients were eligible if they had disease-free survival (DFS) for 5 consecutive years in other malignancies treated by single surgery; Cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  2. Major surgical treatment, open biopsy, or significant traumatic injury within 28 days before the start of study treatment;
  3. Subjects with any severe and/or uncontrolled illness, including:

     1. Patients with ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (including Corrected QT Interval (QTc)≥450ms(male), QTc≥ 470ms(female)) and ≥ grade 2 congestive heart failure (NYHA classification);
     2. Severe active or uncontrolled infection (≥ grade 2 infection according to Common Terminology Criteria for Adverse Events (CTCAE) );
     3. Renal failure requiring hemodialysis or peritoneal dialysis;
* Patients with concomitant diseases that seriously endanger the safety of patients or affect the completion of the study, or patients who are considered to be unsuitable for enrollment for other reasons according to the judgment of the investigators.
* patients with previous treatment with anlotinib hydrochloride capsules or similar vascular endothelial growth factor receptor tyrosine kinase inhibitor (VEGFR-TKI) small molecule drugs, such as vandetanib, Cabozantinib, lenvatinib, sunitinib, or sorafenib, etc.;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally Advanced or Metastatic Radioiodine-Refractory Differentiated Thyroid Carcinoma Patients
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to 3 years.
  The proportion of subjects who achieves a best overall response of complete response (CR) or partial response (PR).
Progression-free Survival (PFS) | Baseline up to 3 years.
  From the first dose to the date of objective disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Disease-control Rate (DCR) | Baseline up to 3 years.
  The proportion of subjects response of CR, PR, or stable disease (SD), subjects achieving SD will be included in the DCR if they maintain SD for ≥4 weeks.
Duration of Response (DOR) | Baseline up to 3 years.
  From the date that CR or PR are first occurred to the date of objective disease progression or death, whichever occurs first.
Overall Survival (OS) | Baseline up to 3 years.
  From randomization to the time of death from any cause.
Adverse event rate | Baseline up to 3 years.
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality